CLINICAL TRIAL: NCT04501185
Title: Comparison of Clinical Results of Two Cementless Femoral Stem
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: United Orthopedic Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 202000226A3
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis, Hip
Keywords: total hip arthroplasty; total hip replacement; femoral stem
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- UTS Stem: The subjects who received UTS Stem in total hip arthroplasty.
  Interventions: Device: total hip arthroplasty
- UTF-reduced Stem: The subjects who received UTF-reduced Stem in total hip arthroplasty.
  Interventions: Device: total hip arthroplasty

INTERVENTIONS:
Device: total hip arthroplasty — The indication for total hip arthroplasty is mainly osteoarthritis.

SUMMARY:
In the present study, two types of cementless femoral stem- UTS Stem and UTF-reduced Stem- were utilized in total hip arthroplasty. Due to the design for proximal femur fixation, both femoral stems could prevent stress shielding around the implant, further preventing osteolysis. The difference between both femoral stems is the length, in which UTS Stem is 20% shorter than UTF-reduced Stem. The clinical outcomes of both femoral stems will be compared. Both femoral stems are expected to have equally good radiologic outcome and clinical performance.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is a common orthopedic procedure aimed at improving joint function and alleviating pain in patients with hip joint degeneration. However, the phenomenon of stress shielding-whereby the mechanical properties of the prosthesis lead to reduced load transmission to the surrounding bone-can compromise long-term outcomes. In particular, uncemented THA designs are susceptible to stress shielding, potentially resulting in bone resorption and implant loosening.

To address this challenge, the study focuses on optimizing femoral stem fixation within the proximal femur in two specific stem designs: the UTS and the UTF reduced stem. These stems are strategically designed to enhance load transfer while minimizing stress shielding effects.

A total of 60 patients who are undergoing total hip arthroplasty at Linkou Chang Gung Memorial Hospital will be recruited, including 30 patients in the "UTS" group and 30 patients in the "UTF-reduced" group.The clinical assessments including Success Rate of prosthesis, Numerical Rating Scale (NRS) for pain, Harris Hip Score (HHS), Medical Outcome Study Short Form-36 (SF-36) and : Dual-energy X-ray absorptiometry (DEXA) scanning for bone mineral density monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who receive total hip arthroplasty with either a UTS femoral stem or a UTF-reduced femoral stem after June, 2020
2. Patients who have not received total hip arthroplasty in the past

Exclusion Criteria:

1. Patients who are unable or unwilling to return for follow-up
2. Patients who suffer from mental disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive total hip arthroplasty with either a UTS femoral stem or a UTF-reduced femoral stem after June, 2020 at Chang Gung Memorial Hospital, Linkou
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Success rate | Duration of 1 year
  Failure is defined as removal or revision of any components as a result of mechanical failure or complications.
  Sucess is defined as implants that are sucessfully implanted without any failure for the duration of 1 year.
  The success rate will be represented as a percentage (%).
Numerical Rating Scale | Change from baseline at 1 year
  Numerical Rating Scale is a patient-reported outcome measure. The scale ranges from 0 to 10. A score of 0 represents no pain, while a score of 10 represents extreme pain.
Harris Hip Score | Change from baseline at 1 year
  Harris Hip Score includes 4 sections that evaluate pain, function, deformity, and range of motion. Total scores is from 0 to 100, higher scores represent a better outcome.
Medical Outcome Study Short Form-36 | Change from baseline at 1 year
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients. It consists of two sections, physical component summary and mental component summary, with 36 items in total.
DEXA scanning | Change from baseline at 1 year
  DEXA scanning is used to monitor and quantify bone mineral density, which helps to understand if the implant has an effect on the change of bone mineral density.

SECONDARY OUTCOMES:
Radiolucent line | Change from baseline at 1 year
  Radiologic analysis helps observe the existence of radiolucent lines, which can be analyzed to determine if implant loosening occurs.
Valgus/Varus alignment | Change from baseline at 1 year
  Radiologic analysis helps measure the degree of the alignment of the hip.
Morphology of the proximal femur | at baseline
  Morphology of the proximal femur was classified using Dorr Type.

CONTACTS AND LOCATIONS:
Overall Officials: Pang-Hsin Hsieh, MD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Joint Reconstruction Division at Chang Gung Memorial Hospital, Linkou, Taoyuan, Taiwan